CLINICAL TRIAL: NCT00867945
Title: Pregnancy-Induced Analgesia - A Longitudinal Study of DNIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Ruth Landau, Professor, University of Washington
Other Study IDs: 35811-A
Record Dates: First submitted 2009-03-20; First posted 2009-03-24 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1. Pregnant Women
- 2. Non-Pregnant Controls
- 3. IVF controls

SUMMARY:
The investigators hypothesize that pregnancy-induced analgesia might be the result of enhanced descending noxious inhibitory activity.

DETAILED DESCRIPTION:
Pregnancy-induced analgesia has been described in several studies (Gintzler 1980; Sander and Gintzler 1987; Jarvis et al. 1997). Obvious mechanisms underlying pregnancy-induced analgesia involve hormonal changes during gestation (Fillingim and Ness 2000). Existing studies during pregnancy and peripartum have focused on standard characteristics of nociception, using non-dynamic quantitative sensory testing such as pain threshold/tolerance or suprathreshold stimuli (Goolkasian and Rimer 1984; Sengupta and Nielsen 1984; Cogan and Spinnato 1986; Dunbar et al. 1988; Whipple et al. 1990; Shapira et al. 1995; Saisto et al. 2001; Bajaj et al. 2002; Carvalho et al. 2006; Ohel et al. 2007), with its relative limitations of studying only the afferent nociceptive input produced in the peripheral nervous system.

The two systems that are of prime importance in pain modulation within the CNS are the inhibitory system (descending noxious inhibitory control (DNIC)) and the excitatory system, with the balance of pain being more heavily influenced by the former (Godfrey and Mackey 2008).

The primary aim of this study is to use psychophysical tests to study both the inhibitory and excitatory pain pathways using the DNIC paradigm and temporal summation longitudinally during pregnancy, compared to an age-matched control group of non-pregnant women.

We added the In Vitro Fertilization (IVF) sub-population to the PIA study to study them as a control group (in addition to studying non-pregnant controls and pregnant women). We are studying this sub population prior to their egg retrieval procedure and a short phone survey with participants post egg-retrieval. If the subject becomes pregnant, we would recruit them to enroll in the PIA pregnant population cohort.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Cohort: Inclusion criteria for participation are (1) women aged between 18 and 45 yr, (2) nulliparous or ASA physical status class I or II women, (3) singleton pregnancy, (4) no more than 14 completed weeks gestational age at the time of enrollment into the study, (5) uncomplicated pregnancy, and (6) delivery planned to be conducted at UW/Stanford University.
* Non-pregnant Control Cohort: Inclusion criteria for participation are (1) women aged between 18 and 45 yr, (2) nulliparous or ASA physical status class I or II women, (3) and not planning on taking oral-contraceptives or carrying a hormonal-coated IUD.

Non-inclusion Criteria:

* Pregnant Cohort: Non-inclusion criteria are (1) multiparous women, (2) non-English speaking women (subjects have to be able to understand the DNIC procedure and answer questionnaires), (3) women unable to understand the concept of VNPS at the time of informed consent (involving mental health issues), (4) a history of anxiety or depression, or chronic consumption of opiates, antidepressants, or anticonvulsants; and (5) intake of opioids, acetaminophen, or NSAIDs 48h prior to the psychophysical test.
* Non-pregnant Control Cohort: Non-inclusion criteria are the same as the Pregnant Cohort as well as (6) irregular menstrual cycles (defined as < 21 days or > 35 days).

Exclusion Criteria:

* Pregnant Cohort: Exclusion criteria is a pregnancy complicated by preeclampsia or preterm delivery (< 37 weeks gestation).
* Non-pregnant Control Cohort: Exclusion criteria is development of irregular cycles.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: maternity clinic - Pregnant Cohort community sample - Non-pregnant Control Cohort
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To use psychophysical tests to study both the inhibitory and excitatory pain pathways using the DNIC paradigm and temporal summation longitudinally during pregnancy, compared to an age-matched control group of non-pregnant women. | Pregnant Cohort - each trimester and postpartum; Control Cohort - twice a menstrual cycle, 4 cycles, over 7 months

SECONDARY OUTCOMES:
Questionnaires, pain scores, amount of analgesics required, overall experience of labor and delivery | Questionnaires - Same as Primary Outcome Measure; other three measures - at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Landau, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - University of Washington, Seattle, Washington